CLINICAL TRIAL: NCT02377219
Title: Bisphenol A Exposure, Ovarian Function and Assisted Reproductive Technology Outcome.
Acronym: FIVPHENOL
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment target not obtained
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: RC31/12/0571; PHRC 2012 (Other Grant/Funding Number: Ministry of Health)
Record Dates: First submitted 2013-12-17; First posted 2015-03-03 (Estimated); Last update posted 2019-07-15 (Actual); Status verified 2019-07

CONDITIONS: Female Reproductive Problem; Male Reproductive Problems
MeSH Terms: interventions — Hematologic Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- couples (Experimental): couples attending an IVF or intra cytoplasmic sperm injection (ICSI) attempt have hormonal and blood analysis
  Interventions: Other: hormonal and blood analysis

INTERVENTIONS:
Other: hormonal and blood analysis

SUMMARY:
Our goal is to prospect the relationships between Bisphenol A (BPA) exposure (measured as its free and conjugated forms in blood and urine) and embryo implantation rate (measured as the ratio between the number of gestational sacs and the number of transferred embryos) after assisted reproductive technology. In order to reduce the confusion factors, the population study is limited to young women (aged 28 to 34), with regular menstrual cycles and without any medical event that could affect the implantation process

DETAILED DESCRIPTION:
Among the various suspected adverse effects of BPA on human health, studies on the possible effects of BPA on reproduction are limited. Animal and in vitro studies indicate that BPA exposure can lead to disrupted oocyte maturation, E2 suppression and early pregnancy loss caused by chromosomal abnormalities. In the woman, studies about the consequences of BPA exposure on reproduction is a very difficult task since gametogenesis in the woman spreads over decades, from the intra-uterine life where meiosis is initiated to the end of the reproductive period at menopause. Recently, a decreased survival of human foetal oocytes cultured in vitro in the presence of BPA has been shown suggesting that in vivo exposure in foetal life could affect the ovarian reserve. Furthermore, a negative association between urinary BPA level and serum peak E2, oocyte yield and blastocyst formation has been suggested on a limited population of women performing ART. These results suggest that, in adulthood, both quantity and quality of human oocytes could be affected by BPA exposures. The study aims to respond to these questions by evaluating the relationships between BPA exposition levels and embryo implantation rates (as a marker of oocyte quality) and anti-Mullerian hormon (AMH) levels (as a marker of ovarian reserve) in large population of young adult women performing ART. BPA exposure will be assessed at two times in both blood and urine: 1°) before the ovarian stimulation at the time of ovarian reserve tests and 2°) at the end of the ovarian stimulation the day of the ovarian puncture for IVF.

ELIGIBILITY:
Inclusion Criteria:

* Couples attending an IVF or ICSI attempt whose woman is aged 28 ans to 34 at inclusion time
* Regular menstrual cycles (between 27 and 33 days)
* 1st or 2nd IVF or ICSI attempt with an embryo transfer at D2 or D3

Exclusion Criteria:

* couple already included in the study
* ovarian surgery history
* uterine (malformation, diethylstilbestrol (DES) syndrome, adenomyosis…) or systemic pathology that can affect implantation (thrombophilia, antiphospholipids syndrome…)
* chemotherapy history for the woman
* any endocrinopathy (except dysthyroid) in the woman
* any pelvic surgery for the woman in the 3 months preceding inclusion
* endometriosis
* ICSI with testicular sperm
* Positive viral load for HIV, hepatitis C virus or hepatitis B virus (HCV or HBV) during the year preceding inclusion in one or both members of the couple

Ages: 28 Years to 34 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 350 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2019-07 (Actual); Study Completion 2019-07 (Actual)

PRIMARY OUTCOMES:
embryo implantation rate | 6 weeks after implantation
  an ultrasonography between the 5th and 7th week after embryo transfer

SECONDARY OUTCOMES:
serum AMH | 4 days after inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Roger LEANDRI, MD, Principal Investigator — University Hospital, Toulouse
Locations (8):
- France (8):
  - University Hospital, Bordeaux
  - CHRU Brest Hôpital Morvan, Service de Médecine de la Reproduction, Brest
  - University Hospital, Dijon
  - University Hospital, Lille
  - CHU Limoges, Centre d'AMP, Limoges
  - University Hospital, Nantes
  - HOSPITAL, Poissy
  - University Hospital, Toulouse

REFERENCES:
- [Background] Corbel T, Gayrard V, Viguie C, Puel S, Lacroix MZ, Toutain PL, Picard-Hagen N. Bisphenol A disposition in the sheep maternal-placental-fetal unit: mechanisms determining fetal internal exposure. Biol Reprod. 2013 Jul 18;89(1):11. doi: 10.1095/biolreprod.112.106369. Print 2013 Jul. PMID 23699389
- [Background] Leandri RD, Gachet A, Pfeffer J, Celebi C, Rives N, Carre-Pigeon F, Kulski O, Mitchell V, Parinaud J. Is intracytoplasmic morphologically selected sperm injection (IMSI) beneficial in the first ART cycle? a multicentric randomized controlled trial. Andrology. 2013 Sep;1(5):692-7. doi: 10.1111/j.2047-2927.2013.00104.x. Epub 2013 Jun 21. PMID 23788532